CLINICAL TRIAL: NCT07311785
Title: Accuracy of Maxillary Fixation Using Custom Plates on Nasal Buttress Only Via Minimally Invasive Approach Versus Custom Plates on Nasal and Zygomatic Buttresses Via Conventional Approach in Orthognathic Surgeries: A Randomized Controlled Trial.
Brief Title: Accuracy of Maxillary Fixation Using Custom Plates on Nasal Buttress Only Via Minimally Invasive Approach Versus Custom Plates on Nasal and Zygomatic Buttresses Via Conventional Approach in Orthognathic Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Hamid Khorshed, oral & maxillofacial surgeon, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Omfs 3-3-19
Record Dates: First submitted 2025-12-03; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Orthognathic Surgery
Keywords: orthognathic; minimally invasive; nasal buttress; custom plate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Maxilla fixation using custom plates on nasal buttress only via minimally invasive approach.
  Interventions: Procedure: minimally invasive maxillary fixation
- control (Active Comparator): Maxilla fixation using custom plates on nasal and zygomatic buttresses via conventional vestibular approach.
  Interventions: Procedure: Maxilla fixation using custom plates on nasal and zygomatic buttresses via conventional vestibular approach.

INTERVENTIONS:
Procedure: minimally invasive maxillary fixation — 3D printed patient specific custom plates minimally invasive maxillary fixation on nasal buttress
  Other Names: 2 plates maxillary fixation
  Arms: intervention
Procedure: Maxilla fixation using custom plates on nasal and zygomatic buttresses via conventional vestibular approach. — 3d printed custom plates fixing maxilla on nasal and zygomatic buttresses via conventional vestibular approach.
  Arms: control

SUMMARY:
The goal of this clinical trial is to evaluate of the accuracy maxilla fixation using custom plates on nasal buttress only via minimally invasive approach versus using custom plates on nasal and zygomatic buttresses via conventional approach. The main question it aims to answer is:

• Is the minimally invasive approach accurate and stable ? Researchers will compare minimally invasive technique to the traditional technique of fixation of the maxilla bone to see if it is as accurate and stable.

Participants will:

* Undergo surgey
* Follow up visits weekly for a month then on a monthly basis for 5 more months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dentofacial disharmony and misalignment requiring bimaxillary orthognathic surgeries.
* Patients with no signs or symptoms of active TMDs.
* Highly motivated patients.

Exclusion Criteria:

* Patients who refused to be included in the research.
* Patients with systemic diseases that may hinder the normal healing process or render the patient not fitting for general anaesthesia.
* Patients with intra-bony lesions or infections that may retard the osteotomy healing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the maxilla fixation on CT compared to preoperative plan assessed by superimposition of preoperative and immediate postoperative scans. | from preoperative plan to immediate postoperative (1 week)
  linear measurement of discrepancy between both scans after superimposition

SECONDARY OUTCOMES:
Stability of maxilla fixation by superimposing preoperative and 6months postoperative CT scans | from enrollment to 6 month postoperative
  linear measurement of discrepancy between both scans after superimposition

IPD SHARING:
Plan to Share IPD: Undecided